CLINICAL TRIAL: NCT03496454
Title: Susceptibility of Gambian Adults to PfSPZ-Challenge Infection in the Controlled Human Malaria Infection Model
Acronym: CHMI-Gambia1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Radboud University Medical Center (Other); Sanaria Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SCC 1529
Record Dates: First submitted 2018-03-29; First posted 2018-04-12 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Malaria
Keywords: malaria; infection; controlled
MeSH Terms: conditions — Malaria; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PfSPZ Challenge (Other): this is a basic sciences protocol designed to study the effect of pre-exposure to Plasmodium falciparum (Pf) on malaria parasite kinetics, clinical symptoms and immunity after Controlled Human Malaria Infection by administration of an injection PfSPZ Challenge in Gambian adults. Based on a well-defined serological profile representing the extremes of current malaria exposure in The Gambia, two cohorts will be identified to study the impact of naturally acquired immunity on susceptibility for a Controlled Human Malaria Infection. The classification as a clinical trial results from the administration of the PfSPZ Challenge to the healthy volunteers
  Interventions: Other: PfSPZ Challenge

INTERVENTIONS:
Other: PfSPZ Challenge — The administration of an injection PfSPZ Challenge in Gambian adults

SUMMARY:
Controlled human malaria infection (CHMI) is an important tool for the assessment of the efficacy of novel malaria vaccines and drugs prior to field trials. CHMI also allows for the evaluation of immunity to malaria and parasite growth rates in vivo and thus allows for the assessment of the natural acquisition and loss of malaria immunity. This may be particularly useful in individuals from endemic areas with changing levels of exposure and immunity to malaria. Thus, CHMI in individuals with prior exposure to malaria could be a valuable tool to accelerate malaria vaccine development and inform malaria control programs of changing immunity levels and related disease presentations. In this trial, the investigators intend to study the effect of pre-exposure to Plasmodium falciparum (Pf) on parasite kinetics, clinical symptoms and immunity after CHMI by PfSPZ Challenge in Gambian adults. Based on a well-defined sero-profile representing the extremes of current malaria exposure in The Gambia, two cohorts will be identified to study the impact of naturally acquired immunity on susceptibility for a Controlled Human Malaria Infection.

DETAILED DESCRIPTION:
The main hypothesis is that cumulative exposure to natural Pf infections, as defined by the antibody profile to a defined panel of Pf antigens, is associated with an increasing pre-patent period and/or a reduced parasite growth rate in the CHMI after PfSPZ Challenge. The Primary objectives are to assess safety of PfSPZ Challenge administration in Gambian adults and to determine parasite kinetics in the CHMI model after PfSPZ Challenge in naturally exposed Gambian adults. The Secondary objective is to analyse humoral and cellular immune responses before and after CHMI in Gambian adults with different serological profiles to a panel of defined Pf-antigens.

The study is a single centre open-label clinical trial. The study population will be adult (aged 18 to 35 years) male, healthy subjects with at least 4 years of secondary school education. A total of 30 individuals will be enrolled to participate in the study; 15 with intense previous and recent exposure to malaria infections and 15 with very limited historic exposure to malaria and no evidence of recent malaria infections.

All participants will be checked for parasitaemia by qPCR before inclusion. Two subsequent negative qPCRs are needed before enrolment in the study to assure the absence of a P.falciparum infection. If one of the participants is not fit to participate in the study, another participant who fulfilled enrolment criteria will be included as replacement. For this purpose, two to four additional participants will be screened as back up. Subsequently, all participants will be subjected to a standard controlled human malaria infection (CHMI) by IV administration of a dose of 3.2 x 10^3 PfSPZ Challenge. After CHMI, participants will be closely followed with regular visits to the clinical trial centre (twice daily until day 15, and daily until day 28 or treatment) consisting of periodic physical examinations, frequent blood sampling and recording of adverse events in their diary. All relevant investigations will be carried out on an outpatient basis, including frequent safety analyses.

Participants should have access to a mobile phone upon which they can be reached 24 hours per day and 7 days per week. As additional safety precaution, participants are required to stay in a hotel/hostel close to the study facility from day 5 post-infection until 3 days after treatment. This mandatory stay in a hotel/hostel is to ensure study participants can be observed at all times and have excellent access to the clinical team. All participants will be treated with a curative regimen of artemether-lumefantrine that radically clears asexual parasites and developing gametocytes. The criteria for treatment post-CHMI will include positive thick smear during follow-up, decision of the study clinician or the local safety monitor, on request of the participant or on day 28 post-CHMI. All participants will be checked for parasites by thick smear at least twice after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males aged ≥ 18 and ≤ 35 years and in good health;
* At least 4 completed years of secondary education;
* Adequate understanding of the procedures of the study in English language;
* Willing (in the investigator's opinion) to comply with all study requirements;
* Willing to complete an informed consent questionnaire and is able to answer all questions correctly;
* Signed written informed consent to participate in the trial;
* Willing to take a course of curative anti-malaria medication;
* Able to communicate well with the investigator and is available to attend all study visits;
* Willing to stay in a hotel close to the trial centre OR willing to be hospitalized in the CSD of MRCG during a part of the study (day 5 post-infection until day 3 after treatment);
* Reachable (24/7) by mobile telephone throughout the entire study period;
* Agrees to refrain from blood donation or for other purposes throughout the study period and after the end of their involvement in the study according to the local blood banking eligibility criteria.
* Agrees to refrain from intensive physical exercise (disproportionate to the participant's usual daily activity or exercise routine) during the malaria challenge period;
* Hb ≥12 g/dl.

Exclusion Criteria:

1. Any history, or evidence at screening, of clinically significant symptoms, physical signs or abnormal laboratory values suggestive of systemic conditions, such as cardiovascular, pulmonary, renal, hepatic, neurological, dermatological, endocrine,malignant, haematological, infectious, immunodeficient, psychiatric and other disorders, which could compromise the health of the participant during the study or interfere with the interpretation of the study results. These include, but are not limited to, any of the following

   1. Body weight <50 kg or Body Mass Index (BMI) <18 or >30 kg/m2 at screening.
   2. A heightened risk of cardiovascular disease, as determined by: an estimated ten year risk of fatal cardiovascular disease of ≥5% at screening, as determined by the Systematic Coronary Risk Evaluation (SCORE); history, or evidence at screening, of clinically significant arrhythmia's, prolonged QT-interval or other clinically relevant ECG abnormalities; or a positive family history of cardiac events in 1st or 2nd degree relatives <50 years old.
   3. A medical history of functional asplenia, G6PD disease or α-thalassaemia disease.
   4. Positive test for sickle cell disease.
   5. History of epilepsy in the period of five years prior to study onset, even if no longer on medication.
   6. Screening tests positive for Human Immunodeficiency Virus (HIV), active Hepatitis B Virus (HBV), Hepatitis C Virus (HCV).
   7. Chronic use of i) immunosuppressive drugs, ii) antibiotics, iii) or other immune modifying drugs within three months prior to study onset (inhaled and topical corticosteroids and oral anti-histamines exempted) or expected use of such during the study period.
   8. Any recent or current systemic therapy with an antibiotic or drug with potential anti-malarial activity (chloroquine, doxycycline, tetracycline, piperaquine, benzodiazepine, flunarizine, fluoxetine, tetracycline, azithromycin, clindamycin, erythromycin, hydroxychloroquine, etc.) (Allowable timeframe for use at the Investigator's discretion).
   9. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years.
   10. Any history of treatment for severe psychiatric disease by a psychiatrist in the past year.
   11. Suspicion or history of drug or alcohol abuse interfering with normal social function in the period of one year prior to study onset.
   12. Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination.
2. qPCR positive for Pf parasites at screening or previous participation in any malaria (vaccine) study.
3. Known hypersensitivity to artemether-lumefantrine.
4. Current use of any drug that is metabolised by the cytochrome enzyme CYP2D6 (e.g. flecainide, metoprolol, imipramine, amitriptyline, clomipramine).
5. Current use of drugs that are known to prolong the QTc interval such as: antiarrhythmics of classes IA and III; neuroleptics and antidepressant agents; certain antibiotics including some agents of the following classes: macrolides, fluoroquinolones, imidazole, and triazole antifungal agents; certain non-sedating antihistaminics (terfenadine, astemizole); cisapride.
6. Disturbances of electrolyte balance, e.g. hypokalaemia.
7. Inability to consume food
8. Use of immunoglobulin or blood products within 3 months prior to enrolment.
9. Participation in any other clinical study in the 30 days prior to the start of the study or during the study period, or prior receipt of an investigational malaria vaccine.
10. Any other condition or situation that would, in the opinion of the investigator, place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol.
11. Any other significant disease, disorder or finding which may significantly increase the risk to the participant because of participation in the study, affect the ability of the participant to participate in the study or impair interpretation of the study data.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Males aged ≥ 18 and ≤ 35 years and in good health
Enrollment: 19 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
frequency and magnitude of adverse events | 28 days
  Frequency, incidence, nature and magnitude of adverse events
time to first detection of parasites and parasites density | 28 days
  to compare time to first detection of parasites and parasite density at first detection by 18S qPCR and varATS qPCR. This time to patency and first parasite density are important indicators of pre-erythrocytic immunity and will be compared between cohorts A and B

SECONDARY OUTCOMES:
Time to Pf-NF54 parasitemia | 28 days
  Time to Pf-NF54 parasitemia after CHMI as assessed by qPCR
parasite growth | day 5 to day 28
  Dynamics of Pf-NF54 parasite growth from day 5 after CHMI until day 28 as assessed by qPCR
differences in immune responses | 28 days
  Intra and inter-group differences in cellular and humoral immune responses

CONTACTS AND LOCATIONS:
Locations (1):
- MRC Unit, Fajara, The Gambia

REFERENCES:
- [Derived] Achan J, Reuling IJ, Yap XZ, Dabira E, Ahmad A, Cox M, Nwakanma D, Tetteh K, Wu L, Bastiaens GJH, Abebe Y, Manoj A, Kaur H, Miura K, Long C, Billingsley PF, Sim BKL, Hoffman SL, Drakeley C, Bousema T, D'Alessandro U. Serologic Markers of Previous Malaria Exposure and Functional Antibodies Inhibiting Parasite Growth Are Associated With Parasite Kinetics Following a Plasmodium falciparum Controlled Human Infection. Clin Infect Dis. 2020 Jun 10;70(12):2544-2552. doi: 10.1093/cid/ciz740. PMID 31402382